CLINICAL TRIAL: NCT03159936
Title: Open Label Phase 2 Pilot Trial of Oral Tofacitinib in Adult Subjects With Discoid Lupus Erythematosus (DLE) and Systemic Lupus Erythematosus (SLE)
Brief Title: Oral Tofacitinib in Adult Subjects With Discoid Lupus Erythematosus (DLE) and Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: unable to identify additional subjects to qualify for enrollment
Sponsor: Tufts Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLE
Record Dates: First submitted 2017-05-02; First posted 2017-05-19 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Discoid Lupus Erythematosus; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Tofacitinib citrate will be administered twice a day starting on Day 1 at the Baseline Visit. Subjects will take one 5 mg tablet by mouth in the morning and one tablet by mouth in the evening for the 6-month study duration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tofacitinib citrate (Experimental): All participants will take one 5 mg tablet by mouth in the morning and one tablet by mouth in the evening for the 6-month study duration.
  Interventions: Biological: Tofacitinib citrate

INTERVENTIONS:
Biological: Tofacitinib citrate — 10 mg daily by mouth
  Other Names: Xeljanz

SUMMARY:
Evaluate the activity and safety of oral tofacitinib in adult patients with discoid lupus erythematosus with or without concurrent SLE.

DETAILED DESCRIPTION:
Discoid Lupus Erythematosus (DLE ) and systemic lupus erythematosus (SLE) can be devastating diseases with a significant impact on quality of life. DLE is currently treated with potent topical steroids, antimalarials, and immunosuppressants. Recent research has determined that DLE is a Th1 mediated disease. There is increasing evidence that JAK inhibitors such as tofacitinib can treat the Th1 mediated diseases such as alopecia areata. Therefore the goal of this study is to determine if JAK inhibitors can successfully treat DLE. Tofacitinib has not previously been studied in DLE. This will be a pilot study that is descriptive for early clinical impressions and molecular mechanisms in order to obtain initial information to potentially design an appropriately -powered phase 2 or 3 study for efficacy of JAK inhibitors that could take place in the future

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years to ≤ 65 years of age with clinical diagnosis of DLE (and at least half of patients with a diagnosis of SLE) as determined by the Principal Investigator by medical history and physical exam.
* Able to understand consent procedure
* Able to comply with protocol activities
* Have had a diagnosis of biopsy proven DLE for at least 6 months prior to Visit 1 (Baseline/Day 1).
* At Screening and Visit 1 (Baseline/Day 1), have had DLE covering at least 5% of total body surface area (BSA) or SLE with DLE covering at least 2% of BSA as determined by the hand print method (one palm is equivalent to 1% BSA).

Exclusion Criteria:

* Patients not able to understand consent procedure
* Patients unable to comply with protocol activities
* Other skin conditions at Baseline that would interfere with evaluation of DLE.
* Topical corticosteroid within the past 2 weeks
* Systemic therapy is allowed if on a stable dose and using for at least 3 months -background therapies outlined in Protocol
* Concomitant use of moderate to potent inhibitors and inducers of CYP3A4/5
* Women who are pregnant or wish to become pregnant, or who are lactating. Women of childbearing potential must use effective contraceptive methods in order to participate in tofacitinib clinical studies
* History of infection requiring hospitalization, parenteral antimicrobial therapy within 6 months prior to first dose of study drug or history of infection requiring antimicrobial therapy within 2 weeks prior to first dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | week 24
  Percent change

CONTACTS AND LOCATIONS:
Overall Officials: David Rosmarin, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No